CLINICAL TRIAL: NCT01822847
Title: Physiological Response of Cortisol to Cardiac Catheterization
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-16583
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Adrenal Insufficiency
Keywords: adrenal; steroids; cortisol; stress
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- catheterization: patients undergoing elective heart catheterization

SUMMARY:
Cortisol is essential for survival. The importance of cortisol response is most apparent in patients with partial or complete deficiency of glucocorticoids during stressful events such as illness or surgery.

DETAILED DESCRIPTION:
It is known that cortisol and other stress hormones increase during acute myocardial infarction as well (9-11). Cardiac catheterization is an essential tool for the management of acute coronary syndrome, and for the evaluation of the burden of coronary artery disease in cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac catheterization, who are willing and able to give consent.

Exclusion Criteria:

* • Patients with .primary or secondary adrenal insufficiency.

  * Patients taking steroids in the doses equivalent of at least 5 mg of prednisone daily for more than 3 weeks in the previous year.
  * Patients undergoing cardiac catheterization in the setting of acute coronary syndrome, eg. STEMI, NSTEMI and unstable angina.
  * Patients with low albumin level (<3.5 g/dL)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 males and females, age 20-90 years who are scheduled for elective cardiac catheterization procedure.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
cortisol change | one month
  On the day of the procedure a total of 4 venous blood samples for random plasma cortisol level will be obtained. Blood will be drawn at 5 minutes prior to the procedure, at 30 minutes and 60 minutes during the cardiac catheterization. Another sample will be drawn in 3 hours after cardiac catheterization prior to the patients discharge. a cortisol level will be drawn at a "nonstressful" visit

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Tarasova, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States